CLINICAL TRIAL: NCT02158884
Title: Patient Response to an Integrated Orthotic and Rehabilitation Initiative for Traumatic Injuries for the Military Treatment Facilities (PRIORITI-MTF)
Brief Title: PRIORITI-MTF Study- Testing Patient Response to the IDEO
Acronym: PRIORITI-MTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-12-2-0032
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2016-12

CONDITIONS: Leg Injuries; Trauma
Keywords: Major extremity trauma; wounded warriors; IDEO; return to run
MeSH Terms: conditions — Leg Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IDEO brace (Other): IDEO brace
  Interventions: Device: IDEO brace

INTERVENTIONS:
Device: IDEO brace — All participants will receive the IDEO brace.
  Other Names: IDEO

SUMMARY:
The goal of the PRIORITI-MTF study is to help determine whether a new type of custom designed brace, called the IDEO ™ along with a physical therapy program, called Return to Run, improves physical function. This brace was developed for wounded warriors who wanted to return to an active lifestyle.

The primary objective of this study is to examine the benefits (and cost-benefits) of an integrated orthotic and rehabilitation program that incorporates the Intrepid Dynamic Exoskeletal Orthosis (IDEO) and the Return to Run (RTR) physical therapy regimen, but designed for scalability in the broader military environment (i.e. beyond San Antonio Military Medical Center where the program was developed)

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60
2. Currently two or more years out from a traumatic unilateral lower extremity injury at or below the knee
3. Healed fractures and able to fully weight bear
4. Evidence of either:

   * Weakness of ankle dorsiflexors and /or plantarflexors resulting from leg injury (defined as less than 4 out of 5 on manual muscle test)
   * Limited ankle dorsiflexion (< 10 degrees) and /or limited ankle plantarflexion (< 20 degrees) resulting from leg injury
   * Mechanical pain with loading to hindfoot/midfoot (>= 50 mm on a 0-100 mm visual analogue scale assessing average daily pain)
   * Ankle or Hindfoot fusion or candidate for ankle or hindfoot fusion
   * Candidate for amputation secondary to ankle/foot impairment

Exclusion Criteria:

1. Ankle plantarflexion or dorsiflexion weakness as a result of spinal cord injury or central nervous system pathology.
2. Non-ambulatory
3. Surgery on study limb anticipated in next 6 months
4. Medical or psychological conditions that would preclude functional testing (ex. severe traumatic brain injury, stroke, renal failure, heart disease, severe anemia)
5. Neurologic, musculoskeletal or other conditions affecting contralateral extremity preventing the study of a healthy control limb
6. Unable or unwilling to participate in two 4-week PT programs
7. Pregnancy
8. Non-English speaking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08-31 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - San Antonio Center for the Intrepid, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 3 military treatment sites in the US.
Pre-assignment Details: Study participants included service members who had functional deficits that interfered with daily activities at least 1 year after a traumatic unilateral lower-extremity injury at or below the knee. This is not a randomized study, all consented participants were provided with an IDEO brace and the Return to Run Physical Therapy program.
Groups:
- IDEO Brace: IDEO brace
  IDEO brace: All participants will receive the IDEO brace and a 4 week integrated "Return to Run" physical therapy program.
Period: Baseline Assessment
Arm/Group | IDEO Brace
Started | 91
Completed | 87
Not Completed | 4
Not completed — Missed performance assessment | 3
Not completed — Missed SMFA | 1
Period: Intervention: IDEO and PT Program
Arm/Group | IDEO Brace
Started | 87
Completed | 81
Not Completed | 6
Not completed — Did not complete PT intervention | 6
Period: Post Intervention (~4 Weeks)
Arm/Group | IDEO Brace
Started | 81
Completed | 71
Not Completed | 10
Not completed — Did not complete performance assessment | 10
Period: 6 Month Assessment
Arm/Group | IDEO Brace
Started (All those that completed the intervention (n = 81) were eligible to start.) | 81
Completed | 61
Not Completed | 20
Not completed — Missed SMFA | 20
Period: 12 Month Assessment
Arm/Group | IDEO Brace
Started (All those that completed the intervention (n = 81) were eligible to start.) | 81
Completed | 64
Not Completed | 17
Not completed — Missed SMFA | 17

BASELINE CHARACTERISTICS:
Population: 87 participants completed baseline assessments; 6 did not complete any of the RTR PT program and were excluded from analysis.
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: As previously noted, only 81 participants completed the RTR PT program.
  years
    number analyzed (Participants) | 81
    (all) | 36.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of the 87 participants that completed baseline assessments, 6 did not complete any of the RTR PT and were excluded from analysis.
  Participants
    number analyzed (Participants) | 81
    Female | 9
    Male | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Of the 87 participants that completed baseline assessments, 6 did not complete any of the RTR PT and were excluded from analysis.
  Participants
    Hispanic: number analyzed (Participants) | 81
    Hispanic | 10
    Non-Hispanic non-white: number analyzed (Participants) | 81
    Non-Hispanic non-white | 15
    Non-Hispanic white: number analyzed (Participants) | 81
    Non-Hispanic white | 54
    Refuse/unknown/missing: number analyzed (Participants) | 81
    Refuse/unknown/missing | 2
Region of Enrollment [Number; unit: participants] — Population: Of the 87 participants that completed baseline assessments, 6 did not complete any of the RTR PT and were excluded from analysis.
  participants
    United States: number analyzed (Participants) | 81
    United States | 81
Self Efficacy for managing a chronic disease 6 item scale [Mean (Standard Deviation); unit: units on a scale] — 6 item scale with observed range of 1-10; score for the full scale is mean of the 6 items. Higher score indicates higher self efficacy. Population: 91 participants were enrolled, 4 did not complete baseline assessments and were withdrawn from the study. An additional 6 received the IDEO but did not complete any of the Return to Run Physical Therapy (RTR PT) sessions and were excluded from analysis.
  units on a scale
    number analyzed (Participants) | 81
    (all) | 38.4 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Four Square Step Test
Description: The 4 step square test is an objective measure of agility. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (This measure is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability).
Time Frame: Baseline
Population: 91 consented at 3 military treatment facilities and received an IDEO. 87 had complete baseline assessments and were included in analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
seconds | 8.0 (2.9)

2. Primary Outcome: Baseline Illinois Agility Test
Description: The Illinois Agility test is an objective measure of agility. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (The Illinois Agility test is part of the "change in functional performance composite measure" calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
seconds | 31.5 (13.7)

3. Primary Outcome: Sit to Stand Test
Description: The Sit to Stand test is an objective measure of strength and power. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (The Sit to Stand test is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)range: > 0 ~ +∞
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
seconds | 10.6 (3.9)

4. Primary Outcome: Timed Stair Assent
Description: The Timed Stair Assent test is an objective measure of strength and power. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (The Timed Stair Assent test is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
seconds | 6.2 (5.3)

5. Primary Outcome: Shuttle Run
Description: The Shuttle run test is an objective measure of agility. It is measured in seconds, with a range of > 0 ~ +∞. Higher values represent better outcomes. (The Shuttle run is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
seconds | 2.5 (1.7)

6. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) Overall Dysfunction (Items 1-34)
Description: The Short Musculoskeletal function Assessment (SMFA) is a participant reported assessment of the impact a musculoskeletal condition on individual function and daily activities. This study used Short Musculoskeletal Function Assessment (SMFA) modules for Overall dysfunction, mobility, daily activities, hand and arm function, and emotional status. Scores range is 0-100. Lower scores indicate better function. Scores are standardized; the formula for standardization is: ((Actual total raw score - lowest possible raw score)/possible raw score range) *100
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 28.6 (13.2)

7. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Mobility
Description: as for outcome 6
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 37.1 (16.6)

8. Primary Outcome: The Short Musculoskeletal Function Assessment (SMFA) - Daily Activities
Description: The Short Musculoskeletal function Assessment (SMFA) is a participant reported assessment of the impact a musculoskeletal condition on individual function and daily activities. This study used Short Musculoskeletal Function Assessment (SMFA) modules for Overall dysfunction, mobility, daily activities, hand and arm function, and emotional status. Scores range is 0-100. Lower scores indicate better function. Scores are standardized; the formula for standardization is ((Actual total raw score - lowest possible raw score)/possible raw score range) *100
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 31.0 (18.3)

9. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Hand and Arm Function
Description: The Short Musculoskeletal function Assessment (SMFA) is a participant reported assessment of the impact a musculoskeletal condition on individual function and daily activities. This study used Short Musculoskeletal Function Assessment (SMFA) modules for Overall dysfunction, mobility, daily activities, hand and arm function, and emotional status. Scores range is 0-100. Lower scores indicate better function. Scores are standardized; the formula for standardization is:
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 2.0 (4.7)

10. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Emotional Status
Description: The Short Musculoskeletal function Assessment (SMFA) is a participant reported assessment of the impact a musculoskeletal condition on individual function and daily activities. This study used Short Musculoskeletal Function Assessment (SMFA) modules for Overall dysfunction, mobility, daily activities, hand and arm function, and emotional status. Scores range is 0-100. Lower scores indicate better function. Scores are standardized; the formula for standardization is: Scores are standardized. The formula for standardization is:
  ((Actual total raw score - lowest possible raw score)/possible raw score range) *100
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 44.4 (20.8)

11. Primary Outcome: Veterans RAND 12 Item Health Survey - Physical Component Summary
Description: The Veterans RAND 12 Item Health Survey (VR-12) is a participant reported global health measure assessing the participant's overall perspective of their health status. Responses are summarized into 2 scores, a Physical Component Score (PCS) (range 0-100) and a Mental Component Score (MCS) (range 0-100). The 12 items correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Higher scores indicate better outcomes.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 32.9 (9.2)

12. Primary Outcome: Veterans RAND 12 Item Health Survey (VR-12) - Mental Health Component Summary
Description: as for outcome 11
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 87
score on a scale | 53.2 (11.7)

13. Primary Outcome: 4 Step Square Test
Description: The 4 step square test is an objective measure of agility. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (This measure is part of the change in functional performance composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)
Time Frame: Post intervention (approx 4 weeks post IDEO fit)
Population: 91 consented at 3 military treatment facilities and received an IDEO. 81 completed the intervention and were included in analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 81
seconds | 6.1 (1.9)

14. Primary Outcome: Illinois Agility Test
Description: The Illinois Agility Test is an objective measure of agility. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (This measure is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability)
Time Frame: Post intervention (approx 4 weeks post IDEO fit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 81
seconds | 22.3 (4.2)

15. Primary Outcome: Sit to Stand Test
Description: The Sit to Stand Test is an objective measure of strength and power. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (This measure is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability).
Time Frame: Post intervention (approx 4 weeks post IDEO fit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 81
seconds | 7.9 (2.1)

16. Primary Outcome: Timed Stair Assent Test
Description: The Timed Stair Assent test is an objective measure of strength and power. It is measured in seconds, with a range of > 0 ~ +∞. Lower values represent better outcomes. (This measure is part of the "change in functional performance" composite measure calculated using the mean of participant's score across several objective performance measures of agility, strength and power, speed, and postural stability).
Time Frame: Post intervention (approx 4 weeks post IDEO fit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IDEO Brace
Number analyzed (Participants) | 81
seconds | 4.2 (1.2)

17. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Overall Dysfunction
Description: as for outcome 6
Time Frame: 6 months
Population: 91 consented at 3 military treatment facilities &received an IDEO (87 had complete baseline assessments). Of the 87, 6 (6.7%) did not participate in RTR PT sessions & were excluded from analysis; of the 81 completing RTR, 10 did not do a performance assessment & 10 missed patient reported outcome surveys leaving 61 in the 6 month analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 24.9 (15.8)

18. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Mobility
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 30.3 (19.2)

19. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Daily Activities
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 25.2 (21.4)

20. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Hand and Arm Function
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 3.2 (7.1)

21. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Emotional Status
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 42.4 (22.7)

22. Primary Outcome: Veterans RAND 12 Item Health Survey (VR-12) - Physical Component Summary (PCS)
Description: as for outcome 11
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 38.6 (10.1)

23. Primary Outcome: Veterans RAND 12 Item Health Survey (VR-12) Mental Health Component Summary (MCS)
Description: as for outcome 11
Time Frame: 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 61
score on a scale | 52.6 (11.0)

24. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Overall Dysfunction
Description: as for outcome 6
Time Frame: 12 months
Population: 91 consented at 3 military treatment facilities and received an IDEO (87 had complete baseline assessments). Of the 87, 6 (6.7%) did not participate in RTR PT sessions & were excluded from analysis; of the 81 completing RTR, 10 missed performance assessment & 7 did not complete patient reported outcome surveys, leaving 64 in the 12 month analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 23.1 (14.3)

25. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Mobility
Description: as for outcome 6
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 28.9 (17.2)

26. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Daily Activities
Description: as for outcome 6
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 23.1 (18.9)

27. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Hand and Arm Function
Description: as for outcome 6
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 3.0 (5.9)

28. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA) - Emotional Status
Description: as for outcome 6
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 39.2 (23.0)

29. Primary Outcome: Veterans RAND 12 Item Health Survey (VR-12) - Physical Component Summary (PCS)
Description: The Veterans RAND 12 Item Health Survey (VR-12) is a participant reported global health measure assessing the participant's overall perspective of their health status. Responses are summarized into 2 scores, a Physical Component Score (PCS) and a Mental Component Score (MCS). Scored on a 5 point Likert scale, the 12 items correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The United States population averages 50 points on both the PCS and MCS (scores may range from 0-100 on each). The United States population standard deviation is 10 points. Higher scores indicate better outcomes.
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 40.1 (11.0)

30. Primary Outcome: Veterans RAND 12 Item Health Survey (VR-12) - Mental Health Component Summary (MCS)
Description: The Veterans RAND 12 Item Health Survey (VR-12) is a participant reported global health measure assessing the participant's overall perspective of their health status. Responses are summarized into 2 scores, a Physical Component Score (PCS) and a Mental Component Score (MCS). Scored on a 5 point Likert scale, the 12 items correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The United States population averages 50 points on both the PCS and MCS (scores may range from 0-100). The United States population standard deviation is 10 points. Higher scores indicate better outcomes.
Time Frame: 12 months
Population: 91 consented at 3 military treatment facilities & received an IDEO (87 had complete baseline assessments). Of the 87, 6 (6.7%) did not participate in RTR PT sessions & were excluded from analysis; of the 81 completing RTR, 10 missed performance assessment & 7 did not complete patient reported outcome surveys, leaving 64 in the 12 month analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEO Brace
Number analyzed (Participants) | 64
score on a scale | 53.5 (10.2)

ADVERSE EVENTS:
Time Frame: Reported quarterly through study completion, approximately 12M.
Arm/Group | IDEO Brace
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT02158884/Prot_SAP_ICF_000.pdf